CLINICAL TRIAL: NCT00461435
Title: Slowing the Degenerative Process, Long Lasting Effect of Hyperbaric Oxygen Therapy in Retinitis Pigmentosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SS01
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Procedure: hyperbaric oxygen therapy

SUMMARY:
Our aim was to assess the role and usefulness of Hyperbaric oxygen therapy in a long lasting period, assessing its efficacy on rescuing retinal photoreceptors and preserving visual function in retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clearly hereditary RP (we performed to all of them genetic analysis for rhodopsin, and peripherin genes, only 4 patient with ADRP showed point mutation 3 on codon 135 and 1 on codon 347); best corrected visual acuity (BCVA) ≥ 0.50 logMAR; visual field ≥ 3 degree diameter circle; recordable ERG.

Exclusion Criteria:

* Exclusion criteria were: patients with sporadic RP; BCVA ≤ 0.50 logMAR; visual field ≤ 3 degree diameter circle; not recordable ERG.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Maria Vingolo, PH.D., Principal Investigator — Policlinico Umberto I, Dipartimento di Oftalmologia
Locations (1):
- Azienda Policlinico Umberto I, Rome, Italy